CLINICAL TRIAL: NCT01078272
Title: The Saint Francis Remote Ischemic Preconditioning Trial (SaFR)
Acronym: SaFR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment inadequate
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Principal Investigator, Nathaniel Reichek MD, Director, Research Department and Cardiac Imaging Program, St. Francis Hospital, New York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-25
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Atherosclerosis; Percutaneous Coronary Intervention; Coronary Stenting; Coronary Stenosis; Remote Ischemic Preconditioning
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote Ischemic Preconditioning (RIPC) (Experimental): Randomized subjects who are treated immediately prior to stenting with remote ischemic preconditioning consisting of 3 5 minute blood pressure cuff inflations to occlude the brachial artery in their nondominant arms, with intervening 5 minute rest periods.
  Interventions: Other: Remote ischemic preconditioning
- Sham Remote Ischemic Preconditioning (Placebo Comparator): Patients who prior to stenting have the RIPC blood pressure cuff placed but not inflated for 3 5 minute episodes with 5 minute rest periods.
  Interventions: Other: Sham Remote Ischemic Preconditioning

INTERVENTIONS:
Other: Remote ischemic preconditioning — Randomized subjects are treated immediately prior to stenting with remote ischemic preconditioning consisting of 3 5 minute blood pressure cuff inflations to occlude the brachial artery in their nondominant arms, with intervening 5 minute rest periods.
  Arms: Remote Ischemic Preconditioning (RIPC)
Other: Sham Remote Ischemic Preconditioning — Randomized subjects who are exposed immediately prior to stenting to sham remote ischemic preconditioning consisting of 3 5 minute blood pressure cuff placements without inflation on their nondominant arms, with intervening 5 minute rest periods.
  Arms: Sham Remote Ischemic Preconditioning

SUMMARY:
This study tests the hypothesis that repeated inflation of a blood pressure cuff on the arm will improve results of coronary stent implantation by:

* reducing chest pain and electrocardiogram changes during balloon inflation to place the stent
* reducing leakage of heart muscle protein(troponin) into the blood stream after stent placement, indicated reduced damage to heart muscle during stent implantation
* increases in molecules in the blood that promote dilation of arteries
* reduced evidence of heart muscle damage on MRI immediately after stenting
* improved patient outcomes over six months with fewer adverse cardiovascular events(heart attack, acute coronary syndrome,renarrowing of the stented artery, heart failure, death, stroke, transient ischemic attack)
* improved heart structure and function at 6 months after stenting

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable chronic coronary artery disease scheduled for elective percutaneous intervention.

Exclusion Criteria:

* Recent (1 month) myocardial infarction
* Acute coronary syndrome
* Chest pain at res
* Estimated glomerular filtration rate(GFR)<45 mL/min/1.73 m2
* Frequent premature atrial or ventricular contractions or atrial fibrillation
* Any contraindication to MRI including implanted non MRI compatible medical devices or ferromagnetic materials such as shrapnel
* Inability to breath-hold
* Severe claustrophobia
* Deafness
* Persistent tremor
* Inability to follow instructions.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
MACE | 6 months post-stenting
  MACE is defined as a combined endpoint including: heart attack, acute coronary syndrome,restenosis of the stented artery, new heart failure stroke, transient ischemic attack or death

SECONDARY OUTCOMES:
troponin I | 24 hours
  prevalence of cTn I > 0.12 nG/ml in active RIPC and placebo groups
chest pain during stenting | immediate during procedure
  compare frequency, severity(1-10 scale) and duration of chest pain during stent implantation
ST segment changes during stent implantation | immediate
  compare prevalence and severity of electrocardiographic ST segment elevation or depression during stent implantation between active and placebo groups
MRI delayed enhancement | 1-7 days after stenting
  Compare prevalence and volume of myocardial delayed gadolinium enhancement in active and placebo groups
Late left ventricular volumes and ejection fraction | 6 months
  Compare left ventricular ejection fraction, end-diastolic and end-systolic volumes between active and placebo groups at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Reichek, MD, Principal Investigator — St. Francis Hospital-The Heart Center, Roslyn, NY
Locations (1):
- St. Francis Hospital-The Heart Center, Roslyn, New York, United States

REFERENCES:
- See also: First randomized trial of RIPC for coronary stenting — http://www.ncbi.nlm.nih.gov/pubmed/19188504?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=39
- See also: editorial review of remote ischemic preconditioning in coronary disease — http://www.ncbi.nlm.nih.gov/pubmed/19221230?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=37